CLINICAL TRIAL: NCT06136039
Title: Effect of Sarcopenia on Clinical Outcome of Total Knee Arthroplasty
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Byungwoo Cho, Clinical Associate professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3-2022-0137
Record Dates: First submitted 2023-11-10; First posted 2023-11-18 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: This study has prospective cohort design. Prior to surgery, a sarcopenia assessment was conducted to categorize patients into sarcopenia and normal groups. Sarcopenia was reassessed at 6 and 12 months post-surgery for comparison with the preoperative state. Additionally, clinical outcomes of patients were evaluated at 3, 6, and 12 months post-surgery for comparison between the normal and sarcopenia groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sarcopenia (Experimental): Patients were categorized into preoperative sarcopenia
  Interventions: Procedure: Arm I (Sarcopenia); Procedure: Arm II(Normal)
- normal (No Intervention): normal groups according to the AWGS 2019 criteria.

INTERVENTIONS:
Procedure: Arm I (Sarcopenia) — Same as standard treatment
  Arms: Sarcopenia
Procedure: Arm II(Normal) — Same as standard treatment
  Arms: Sarcopenia

SUMMARY:
As human life expectancy increases, the prevalence of degenerative osteoarthritis of the knee joints is steadily rising, leading to a significant surge in the frequency of total knee arthroplasty (TKA). However, research on sarcopenia in the population that comprises the primary recipients of these orthopedic joint surgeries has been notably lacking. Since the release of the 2019 Consensus update on sarcopenia by the Asian Walking Group for Sarcopenia (AWGS) in 2020, research on sarcopenia has gained momentum in various domains. Yet, as previously mentioned, the field of orthopedics still lags behind in investigating sarcopenia. Therefore, it is believed that establishing the relationship between sarcopenia and surgical outcomes in the elderly, who are the primary targets of orthopedic joint replacement surgery, could offer insights to further enhance the results of joint replacement surgeries.

ELIGIBILITY:
Inclusion Criteria:

* A woman aged 60 or older who is undergoing TKA due to degenerative osteoarthritis of the knee joint at the our institution.

Exclusion Criteria:

1. Male
2. Under 60 years of age
3. Patients with a history of rheumatoid arthritis, traumatic joint disease, and post-infection joint disease
4. Patients who cannot undergo tests for muscle weakness diagnosis A. Patients unable to walk B. Patients unable to stand alone due to conditions like cerebral palsy or brain disorders C. Patients unable to use muscle strength
5. Patients considered inappropriate for recruitment in this study based on the judgment of the research team.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
handgrip strength, gait speed, SPPB, ASM) | 6, 12months after surgery
  Handgrip strengths were measured using a handgrip dynamometer before surgery. low muscle mass AND (low physical performance OR low strength) : sarcopenia low muscle mass AND (low physical performance AND low strength) : severe sarcopenia
gait speed | 6, 12months after surgery
  Gait speed was measured using a dedicated camera equipped with LiDAR sensors.
SPPB | 6, 12months after surgery
  The Short Physical Performance Battery was measured using a dedicated device that included a force plate.
ASM | 6, 12months after surgery
  Appendicular Skeletal Muscle Mass was measured through Bioelectrical Impedance Analysis.

SECONDARY OUTCOMES:
Knee Society Score | 3, 6, and 12months after surgery
  The original KSS has a "Knee Score" section (7 items) and a "Functional Score" section (3 items). Both sections are scored from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions
WOMAC | 3, 6, and 12months after surgery
  Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC measures five items for pain (score range 0-20), two for stiffness (score range 0-8), and 17 for functional limitation (score range 0-68).
EQ-5D | 3, 6, and 12months after surgery
  The EuroQol 5 Dimension (EQ-5D) is a self-report survey that measures quality of life across 5 domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression
UCLA score | 3, 6, and 12months after surgery
  The UCLA Activity Scale (UCLA) is a questionnaire assessing physical activity level from 1 (low) to 10 (high) in patients undergoing hip or knee arthroplasty

CONTACTS AND LOCATIONS:
Locations (1):
- GangnamSeverance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen LK, Woo J, Assantachai P, Auyeung TW, Chou MY, Iijima K, Jang HC, Kang L, Kim M, Kim S, Kojima T, Kuzuya M, Lee JSW, Lee SY, Lee WJ, Lee Y, Liang CK, Lim JY, Lim WS, Peng LN, Sugimoto K, Tanaka T, Won CW, Yamada M, Zhang T, Akishita M, Arai H. Asian Working Group for Sarcopenia: 2019 Consensus Update on Sarcopenia Diagnosis and Treatment. J Am Med Dir Assoc. 2020 Mar;21(3):300-307.e2. doi: 10.1016/j.jamda.2019.12.012. Epub 2020 Feb 4. PMID 32033882
- [Background] Lopez de la Oliva AR, Campos-Sandoval JA, Gomez-Garcia MC, Cardona C, Martin-Rufian M, Sialana FJ, Castilla L, Bae N, Lobo C, Penalver A, Garcia-Frutos M, Carro D, Enrique V, Paz JC, Mirmira RG, Gutierrez A, Alonso FJ, Segura JA, Mates JM, Lubec G, Marquez J. Author Correction: Nuclear Translocation of Glutaminase GLS2 in Human Cancer Cells Associates with Proliferation Arrest and Differentiation. Sci Rep. 2021 Jan 4;11(1):249. doi: 10.1038/s41598-020-80651-0. No abstract available. PMID 33397990
- [Background] Pichonnaz C, Bassin JP, Currat D, Martin E, Jolles BM. Bioimpedance for oedema evaluation after total knee arthroplasty. Physiother Res Int. 2013 Sep;18(3):140-7. doi: 10.1002/pri.1540. Epub 2012 Nov 27. PMID 23188719
- [Background] Wagner DR. Case study: Effect of surgical metal implant on single frequency bioelectrical impedance measures of an athlete. Physiol Rep. 2020 Jun;8(11):e14464. doi: 10.14814/phy2.14464. PMID 32472735
- [Background] Ardeljan AD, Polisetty TS, Palmer J, Vakharia RM, Roche MW. Comparative Analysis on the Effects of Sarcopenia following Primary Total Knee Arthroplasty: A Retrospective Matched-Control Analysis. J Knee Surg. 2022 Jan;35(2):128-134. doi: 10.1055/s-0040-1713355. Epub 2020 Jul 6. PMID 32629511
- [Background] Babu JM, Kalagara S, Durand W, Antoci V, Deren ME, Cohen E. Sarcopenia as a Risk Factor for Prosthetic Infection After Total Hip or Knee Arthroplasty. J Arthroplasty. 2019 Jan;34(1):116-122. doi: 10.1016/j.arth.2018.09.037. Epub 2018 Sep 20. PMID 30337254
- [Background] Liao CD, Chen HC, Huang SW, Liou TH. Impact of sarcopenia on rehabilitation outcomes after total knee replacement in older adults with knee osteoarthritis. Ther Adv Musculoskelet Dis. 2021 Mar 12;13:1759720X21998508. doi: 10.1177/1759720X21998508. eCollection 2021. PMID 33786069
- [Background] Shin KY, Park KK, Moon SH, Yang IH, Choi HJ, Lee WS. Vitamin D deficiency adversely affects early post-operative functional outcomes after total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2017 Nov;25(11):3424-3430. doi: 10.1007/s00167-016-4209-8. Epub 2016 Jun 17. PMID 27316697
- [Derived] Lee WS, Park KK, Kwon HM, Park JY, Kim TH, Cho BW. A prospective, single-center longitudinal study on the operational definition of sarcopenia in patients undergoing total knee arthroplasty. Eur Geriatr Med. 2025 Nov 28. doi: 10.1007/s41999-025-01368-9. Online ahead of print. PMID 41313412